CLINICAL TRIAL: NCT04884555
Title: Association of Extracellular Thiol-disulfide and Intracellular Oxidized-reduced Glutathione Homeostasis With Severity and Clinical Prognosis of Post-stroke Patients
Brief Title: SH-SS and GSH-GSSG Homeostasis in Post-stroke Patients
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Other Study IDs: AIBU-FTR-TA-01
Record Dates: First submitted 2021-04-21; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Stroke
Keywords: stroke; Thiol; Disulphide; Glutathione
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post-stroke patient: patients with subacute stroke who have a stroke for the first time and admitted to the hospital for the first rehabilitation treatments
  Interventions: Other: Standard neurorehabilitation; Diagnostic Test: Thiol-Disulphide Homeostasis; Diagnostic Test: Oxidized-reduced Glutathione Homeostasis
- Control: healthy volunteers who have not got any known disease and any sign in physical examination
  Interventions: Diagnostic Test: Thiol-Disulphide Homeostasis; Diagnostic Test: Oxidized-reduced Glutathione Homeostasis

INTERVENTIONS:
Other: Standard neurorehabilitation — Routine post-stroke rehabilitation
  Groups: post-stroke patient
Diagnostic Test: Thiol-Disulphide Homeostasis — Monitoring the levels of thiol and disulphide in serum
Diagnostic Test: Oxidized-reduced Glutathione Homeostasis — Monitoring the levels of intracellular oxidized glutathione and reduced glutathione in whole blood samples

SUMMARY:
In patients undergoing physical therapy after stroke, extracellular thiol-disulfide balance and intracellular oxidized-reduced glutathione balance levels will be monitored. The main objectives of this study are; (1) to determine the differences between thiol-disulfide and GSH-GSSG balances in stroke patients compared to healthy volunteers, (2) to evaluate the relationship of these balances with the severity of stroke, (3) to determine the predictive value of the levels of these balances on clinical prognosis and functional recovery outcomes, and (4) to investigate and to examine the effects of the physical therapy process on these parameters and functional recovery and their relationship with each other.

DETAILED DESCRIPTION:
Stroke is among the most common causes of all deaths and Disability-Adjusted Life Years (DALYs) in the world. There is a close relationship between stroke pathophysiology and post-stroke clinic with oxidative stress. Thiol-disulfide homeostasis systems, which is one of the important extracellular and intracellular oxidative stress markers, showing antioxidant capacity with SH form, and oxidative status with disulfide (SS) form. In this study, we aimed to evaluate the relationship between the clinical outcome of subacute stroke patients and extracellular thiol-disulfide (SH-SS) and intracellular oxidized-reduced glutathione (GSSG-GSH) homeostasis and the comparison of these with healthy volunteers. In addition, the effect of the rehabilitation program on these oxidative stress markers and clinical scores and the predictive value of these oxidative stress parameters on prognosis were also evaluated. The main objectives of this study are; (1) to determine the differences between thiol-disulfide and GSH-GSSG balances in stroke patients compared to healthy volunteers, (2) to evaluate the relationship of these balances with the severity of stroke, (3) to determine the predictive value of the levels of these balances on clinical prognosis and functional recovery outcomes, and (4) to investigate and to examine the effects of the physical therapy process on these parameters and functional recovery and their relationship with each other.

In this study, which is designed as a prospective observational study, patients with subacute stroke who have a stroke for the first time and are admitted to the hospital for the first rehabilitation treatment and healthy volunteers (control group) will be included. The clinical conditions of the patients will be evaluated at the beginning and after the 4-week rehabilitation program at the time of discharge by National Institutes of Health Stroke Scale Scores (NIHSS), modified Rankin Scale (mRS) and Barthel Daily Living Activities Index (BI). Serum and whole blood samples will be obtained from the patient group at the beginning and at discharge, and from the control group. The SH-SS homeostasis parameters (SH, Total SH, SS and SS / SH percent ratio) from serum samples and GSSG-GSH homeostasis parameters (GSH, Total GSH, GSSG and GSSG / GSH percentage ratio) from whole blood samples will be determined. Age, gender, hemiplegic side, type of stroke will be noted. Later, statistical analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a first-ever stroke verified by computed tomography (CT) or magnetic resonance imaging (MRI) reports
* admitted to the hospital for standard neurorehabilitation within 1 to 6 months of stroke onset
* healthy individuals (for control group)

Exclusion Criteria:

* significant acute medical illness (e.g., autoimmune disease, infection, tumor, heart failure, renal or liver dysfunction)
* significant acute neurological illness other than stroke (e.g., head trauma, brain abscess, brain tumor, migraine attack, seizure)
* cannot adapt to work
* previous history of neurorehabilitation therapy
* taking the antioxidant supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-stroke patients group admitted to hospital to take rehablititation and physiotherapy within 1 to 6 months of stroke onset.
  Healthy adult volunteers (control) group (> 18 years of age) with no known disease and no findings on physical examination
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
NIHSS Scores | at baseline (pre-treatment)
  National Institutes Of Health Stroke Scale Scores
NIHSS Scores | after 4 weeks of treatment (post-treatment)
  National Institutes Of Health Stroke Scale Scores
mRS | at baseline (pre-treatment)
  modified Rankin Scales
mRS | after 4 weeks of treatment (post-treatment)
  modified Rankin Scales
BI | at baseline (pre-treatment)
  Barthel Index for Activities of Daily Living
BI | after 4 weeks of treatment (post-treatment)
  Barthel Index for Activities of Daily Living

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Alisik, MD, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brott T, Adams HP Jr, Olinger CP, Marler JR, Barsan WG, Biller J, Spilker J, Holleran R, Eberle R, Hertzberg V, et al. Measurements of acute cerebral infarction: a clinical examination scale. Stroke. 1989 Jul;20(7):864-70. doi: 10.1161/01.str.20.7.864. PMID 2749846
- [Background] Kucukdeveci AA, Yavuzer G, Tennant A, Suldur N, Sonel B, Arasil T. Adaptation of the modified Barthel Index for use in physical medicine and rehabilitation in Turkey. Scand J Rehabil Med. 2000 Jun;32(2):87-92. PMID 10853723
- [Background] Broderick JP, Adeoye O, Elm J. Evolution of the Modified Rankin Scale and Its Use in Future Stroke Trials. Stroke. 2017 Jul;48(7):2007-2012. doi: 10.1161/STROKEAHA.117.017866. Epub 2017 Jun 16. No abstract available. PMID 28626052
- [Background] Erel O, Neselioglu S. A novel and automated assay for thiol/disulphide homeostasis. Clin Biochem. 2014 Dec;47(18):326-32. doi: 10.1016/j.clinbiochem.2014.09.026. Epub 2014 Oct 7. PMID 25304913
- [Background] Alisik, M., Neselioglu, S., & Erel, O. (2019). A colorimetric method to measure oxidized, reduced and total glutathione levels in erythrocytes, Journal of Laboratory Medicine, 43(5), 269-277